CLINICAL TRIAL: NCT01630499
Title: Preventing Breast Cancer Recurrence Through a Tailored Lifestyle Intervention.
Brief Title: My Lifestyle Intervention of Food and Exercise
Acronym: MyLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MyLIFE2012; 427-2012 (Other: UF IRB 01)
Record Dates: First submitted 2012-06-22; First posted 2012-06-28 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast cancer; Breast cancer prevention; Breast cancer recurrence; Weight loss; Weight management; Overweight; Obesity
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Weight Loss; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Lifestyle Intervention (TLI) (Experimental): Participants randomized to the TLI condition will receive a 3-month weight management program tailored to the specific needs of women in remission from breast cancer.
  Interventions: Behavioral: Tailored Lifestyle Intervention (TLI)
- Commercial Weight Loss Program (CLWP) (Active Comparator): Participants randomized to the CWLP condition will receive a 3-month commercial weight loss program (i.e., Weight Watchers) at no cost.
  Interventions: Behavioral: Commercial Weight Loss Program (CWLP)

INTERVENTIONS:
Behavioral: Tailored Lifestyle Intervention (TLI) — The intervention is a nutrition, physical activity, and behavioral weight management program that is tailored to the specific needs of breast cancer survivors.
  Arms: Tailored Lifestyle Intervention (TLI)
Behavioral: Commercial Weight Loss Program (CWLP) — This intervention is a generic, widely-available weight management program.
  Arms: Commercial Weight Loss Program (CLWP)

SUMMARY:
Breast cancer risk, and risk of related health problems (e.g., heart disease), is highest among women with a history of breast cancer (stages 1-3) who are also overweight or obese. The purpose of this study is to compare a tailored nutrition, physical activity, and behavioral weight management program for breast cancer survivors against a widely available commercial weight management program. We hypothesize that an intervention tailored to the unique psychological, nutritional and physical needs of breast cancer survivors will provide superior physiological and psychological benefits compared to an existing commercial program.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21 to 65
* History of stage 1, 2, or 3 breast cancer
* Completed primary treatments (chemotherapy, radiation, and/or surgical treatment) for breast cancer (with or without maintenance therapy) within the last 3 months to 5 years of providing consent
* Be willing/able to attend groups and assessments in Gainesville or Jacksonville
* BMI of 27 to 45 kg/m2
* Weight-stable, i.e., not lost/gained ≥ 10 lbs in the preceding 6 months, or since the end of primary treatment

Exclusion Criteria:

* History of bariatric surgery
* Pregnant, lactating, or planning on becoming pregnant in next 12 months.
* Irritable bowel syndrome
* Serious infectious disease
* Chronic malabsorption syndrome
* Uncontrolled angina within the past 6 months
* History of musculo-skeletal or chronic lung diseases that limit physical activity
* Serum creatinin > 1.5 mg/dL
* Uncontrolled or insulin-dependent diabetes (i.e., hemoglobin A1c< 10 g/dL, fasting serum triglycerides > 400 mg/dL; oral medications are not exclusionary)
* At-rest blood pressure > 140/90 mg/Hg
* Myocardial infarction
* Stroke
* Congestive heart failure
* Chronic hepatitis
* Cirrhosis
* Chronic pancreatitis
* History of solid organ transplantation
* Cancer treatment within past 5 years (other than for breast cancer)
* Any other physical condition (other than history of breast cancer) deemed likely to limit 5-year life expectancy or significantly interfere with individuals' ability to participate in a lifestyle intervention involving eating and physical activity changes.
* Use of antipsychotic medications, monoamine oxidase inhibitors, systemic corticosteroids, human immunodeficiency virus or tuberculosis antibiotics, chemotherapeutics medications, or weight-loss medications.
* Significant psychiatric disorder
* Illicit drug use or excessive use of alcohol (i.e., > 2 drinks/day)
* Currently participating in Weight Watcher's or another weight loss program
* Currently participating in another research study
* Unable to read English at the 5th grade level
* Unable/unwilling to provide informed consent
* Unwilling to receive random assignment to TLI or CWLP

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-10; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline to post-intervention | baseline (month 0), post-intervention (month 3)
Change in body weight from post-intervention to follow-up | post-intervention (month 3), follow-up (month 9)

SECONDARY OUTCOMES:
Change in inflammatory/metabolic disease markers associated with breast cancer recurrence from baseline to post-intervention | baseline (month 0), post-intervention (month 3)
Change in HDL Cholesterol from baseline to post-intervention | baseline (month 0), post-intervention (month 3)
Change in blood glucose control from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  HgA1c and fasting glucose to assess blood glucose control
Change in caloric intake from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  National Cancer Institute's Automated Self-Administered 24-hour recall system (ASA-24)will be utilized to assess dietary intake.
Change in body composition from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Body composition will be assessed using air displacement plethysmography (Bodpod, COSMED, Inc).
Change in waist circumference from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Waist circumference will be measured in triplicate at the top of the iliac crest using a tension controlled tape measure upon exhalation.
Change in sagittal abdominal diameter from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Sagittal abdominal diameter will be measured in triplicate using a Holtain Kahn caliper at the top of the iliac crest upon exhalation.
Change in physical activity from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Physical activity will be assessed using both objective measurement (via triaxial accelerometer) and subjective assessment (via the International Physical Activity Questionnaire, or IPAQ).
Change in health-related quality of life from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Health-related quality of life will be assessed using the European Organization of Research and Treatment of Cancer - Quality of Life (QLQ-30) and the breast-cancer specific addendum (BR-23).
Change in self-efficacy from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
  Self-efficacy to abstain from eating in a variety of situations will be assessed using the Weight Efficacy Lifestyle (WEL) questionnaire.
Use of weight management strategies | post-intervention (month 3)
  The frequency of participants' utilization of specific weight management strategies will be assessed using the Weight Management Questionnaire (WMQ).
Height | baseline (month 0)
  Height will be assessed in order to determine BMI.
Change in blood pressure from baseline to post-intervention. | post-intervention (month 3), follow-up (month 9)
  Systolic and diastolic blood pressure will be assessed at each time point using an appropriately sized cuff after the participant has been sitting quietly for at least 10 minutes.
Change in LDL cholesterol at from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
Change in total cholesterol from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
Change in triglycerides from baseline to post-intervention. | baseline (month 0), post-intervention (month 3)
Change in inflammatory/metabolic disease markers associated with breast cancer recurrence from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
Change in HDL Cholesterol from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
Change in blood glucose control from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
Change in caloric intake from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  National Cancer Institute's Automated Self-Administered 24-hour recall system (ASA-24)will be utilized to assess dietary intake.
Change in body composition from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Body composition will be assessed using air displacement plethysmography (Bodpod, COSMED, Inc).
Change in waist circumference from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Waist circumference will be measured in triplicate at the top of the iliac crest using a tension controlled tape measure upon exhalation.
Change in sagittal abdominal diameter from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Sagittal abdominal diameter will be measured in triplicate using a Holtain Kahn caliper at the top of the iliac crest upon exhalation.
Change in physical activity from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Physical activity will be assessed using both objective measurement (via triaxial accelerometer) and subjective assessment (via the International Physical Activity Questionnaire, or IPAQ).
Change in health-related quality of life from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Health-related quality of life will be assessed using the European Organization of Research and Treatment of Cancer - Quality of Life (QLQ-30) and the breast-cancer specific addendum (BR-23).
Change in self-efficacy from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Self-efficacy to abstain from eating in a variety of situations will be assessed using the Weight Efficacy Lifestyle (WEL) questionnaire.
Use of weight management strategies at follow-up. | follow-up (month 9)
  The frequency of participants' utilization of specific weight management strategies will be assessed using the Weight Management Questionnaire (WMQ).
Change in blood pressure from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
  Systolic and diastolic blood pressure will be assessed at each time point using an appropriately sized cuff after the participant has been sitting quietly for at least 10 minutes.
Change in LDL cholesterol at from post-intervention follow-up | post-intervention (month 3), follow-up (month 9)
Change in total cholesterol from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)
Change in triglycerides from post-intervention to follow-up. | post-intervention (month 3), follow-up (month 9)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mathews, PhD, RD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of North Florida, Jacksonville, Florida

REFERENCES:
- [Background] Pharoah PD, Day NE, Duffy S, Easton DF, Ponder BA. Family history and the risk of breast cancer: a systematic review and meta-analysis. Int J Cancer. 1997 May 29;71(5):800-9. doi: 10.1002/(sici)1097-0215(19970529)71:53.0.co;2-b. PMID 9180149
- [Background] McTiernan A. Behavioral risk factors in breast cancer: can risk be modified? Oncologist. 2003;8(4):326-34. doi: 10.1634/theoncologist.8-4-326. PMID 12897329
- [Background] King MC, Marks JH, Mandell JB; New York Breast Cancer Study Group. Breast and ovarian cancer risks due to inherited mutations in BRCA1 and BRCA2. Science. 2003 Oct 24;302(5645):643-6. doi: 10.1126/science.1088759. PMID 14576434
- [Background] Calle EE, Rodriguez C, Walker-Thurmond K, Thun MJ. Overweight, obesity, and mortality from cancer in a prospectively studied cohort of U.S. adults. N Engl J Med. 2003 Apr 24;348(17):1625-38. doi: 10.1056/NEJMoa021423. PMID 12711737
- [Background] Berclaz G, Li S, Price KN, Coates AS, Castiglione-Gertsch M, Rudenstam CM, Holmberg SB, Lindtner J, Erien D, Collins J, Snyder R, Thurlimann B, Fey MF, Mendiola C, Werner ID, Simoncini E, Crivellari D, Gelber RD, Goldhirsch A; International Breast Cancer Study Group. Body mass index as a prognostic feature in operable breast cancer: the International Breast Cancer Study Group experience. Ann Oncol. 2004 Jun;15(6):875-84. doi: 10.1093/annonc/mdh222. PMID 15151943
- [Background] Nichols HB, Trentham-Dietz A, Egan KM, Titus-Ernstoff L, Holmes MD, Bersch AJ, Holick CN, Hampton JM, Stampfer MJ, Willett WC, Newcomb PA. Body mass index before and after breast cancer diagnosis: associations with all-cause, breast cancer, and cardiovascular disease mortality. Cancer Epidemiol Biomarkers Prev. 2009 May;18(5):1403-9. doi: 10.1158/1055-9965.EPI-08-1094. Epub 2009 Apr 14. PMID 19366908
- [Background] Gallicchio L, Kalesan B, Hoffman SC, Helzlsouer KJ. Non-cancer adverse health conditions and perceived health and function among cancer survivors participating in a community-based cohort study in Washington County, Maryland. J Cancer Surviv. 2008 Mar;2(1):12-9. doi: 10.1007/s11764-008-0046-1. Epub 2008 Feb 12. PMID 18648983
- [Background] Fossa SD, Vassilopoulou-Sellin R, Dahl AA. Long term physical sequelae after adult-onset cancer. J Cancer Surviv. 2008 Mar;2(1):3-11. doi: 10.1007/s11764-007-0039-5. Epub 2007 Dec 4. PMID 18648982
- [Background] Chen Z, Maricic M, Bassford TL, Pettinger M, Ritenbaugh C, Lopez AM, Barad DH, Gass M, Leboff MS. Fracture risk among breast cancer survivors: results from the Women's Health Initiative Observational Study. Arch Intern Med. 2005 Mar 14;165(5):552-8. doi: 10.1001/archinte.165.5.552. PMID 15767532
- [Background] Coups EJ, Ostroff JS. A population-based estimate of the prevalence of behavioral risk factors among adult cancer survivors and noncancer controls. Prev Med. 2005 Jun;40(6):702-11. doi: 10.1016/j.ypmed.2004.09.011. PMID 15850868
- [Background] Bellizzi KM, Rowland JH, Jeffery DD, McNeel T. Health behaviors of cancer survivors: examining opportunities for cancer control intervention. J Clin Oncol. 2005 Dec 1;23(34):8884-93. doi: 10.1200/JCO.2005.02.2343. PMID 16314649
- [Background] Robien K, Demark-Wahnefried W, Rock CL. Evidence-based nutrition guidelines for cancer survivors: current guidelines, knowledge gaps, and future research directions. J Am Diet Assoc. 2011 Mar;111(3):368-75. doi: 10.1016/j.jada.2010.11.014. No abstract available. PMID 21338735
- [Background] Coussens LM, Werb Z. Inflammation and cancer. Nature. 2002 Dec 19-26;420(6917):860-7. doi: 10.1038/nature01322. PMID 12490959
- [Background] Shacter E, Weitzman SA. Chronic inflammation and cancer. Oncology (Williston Park). 2002 Feb;16(2):217-26, 229; discussion 230-2. PMID 11866137
- [Background] Flegal KM, Carroll MD, Ogden CL, Curtin LR. Prevalence and trends in obesity among US adults, 1999-2008. JAMA. 2010 Jan 20;303(3):235-41. doi: 10.1001/jama.2009.2014. Epub 2010 Jan 13. PMID 20071471
- [Background] Vance V, Mourtzakis M, McCargar L, Hanning R. Weight gain in breast cancer survivors: prevalence, pattern and health consequences. Obes Rev. 2011 Apr;12(4):282-94. doi: 10.1111/j.1467-789X.2010.00805.x. Epub 2010 Sep 29. PMID 20880127